CLINICAL TRIAL: NCT00844337
Title: Safety and Efficacy of Simplified Antibiotic Regimens for Outpatient Treatment of Suspected Sepsis in Neonates and Young Infants in Bangladesh
Brief Title: Simplified Antibiotic Regimens for Outpatient Treatment of Suspected Sepsis in Neonates and Young Infants in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Dhaka Shishu Hospital (Other)
Responsible Party: Principal Investigator, Abdullah Baqui, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JHU IRB 1440; USAID GHS-A-00-09-00004-00 (Other Grant/Funding Number: USAID 106744)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Sepsis
Keywords: antibiotic regimens; sepsis; young infants; Bangladeshi; outpatient treatment; Suspected sepsis in young infants
MeSH Terms: conditions — Sepsis | interventions — Gentamicins; Amoxicillin; Penicillins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): One study arm will receive injectable gentamicin once daily and oral amoxicillin twice daily for seven days by comparison to other study arms.
  Interventions: Drug: Gentamicin & Amoxicillin x 7days
- 2 (Active Comparator): Injectable penicillin and gentamicin once daily for two days followed by oral amoxicillin twice daily for five days
  Interventions: Drug: Penicillin & gentamicin x 2 d + Amoxicillin X 5 d
- 3 (Active Comparator): Injectable procaine-benzyl penicillin and gentamicin once daily each for seven days (COMPARISON ARM)
  Interventions: Drug: Standard reference therapy

INTERVENTIONS:
Drug: Gentamicin & Amoxicillin x 7days — Injectable gentamicin once daily and oral amoxicillin twice daily for seven days.
  The dose for gentamicin is 4 - 5 mg/kg/24 hours. The dose for amoxicillin is 90-115 mg/kg/day.
  Other Names: Gentamicin & Amoxicillin
  Arms: 1
Drug: Penicillin & gentamicin x 2 d + Amoxicillin X 5 d — Injectable penicillin and gentamicin once daily for two days followed by oral amoxicillin twice daily for five days. The dose for penicillin is 40,000 - 50,000 U/kg/24 hours, the dose for gentamicin is 4 - 5 mg/kg/24 hours, and the dose for amoxicillin is 90-115 mg/kg/day.
  Other Names: Penicillin; Gentamicin
  Arms: 2
Drug: Standard reference therapy — Injectable procaine-benzyl penicillin and gentamicin once daily each for seven days. The penicillin dose is 40,000 - 50,000 U/kg/24 hours, and the gentamicin dose is 4 - 5 mg/kg/24 hours.
  Arms: 3

SUMMARY:
The primary aim is to establish the non-inferiority of several simplified, home-based antibiotic regimens compared to the standard course of parenteral antibiotics for the empiric treatment of suspected sepsis in Bangladeshi young infants whose parents refuse hospitalization. Three alternative regimens will be compared with a standard (reference) regimen of injectable procaine-benzyl penicillin and gentamicin once daily each for seven days. Alternative regimens are (1) injectable gentamicin once daily and oral amoxicillin twice daily for seven days; (2) injectable penicillin and gentamicin once daily for two days followed by oral amoxicillin twice daily for five days; and (3) injectable gentamicin once daily and oral amoxicillin twice daily for two days followed by oral amoxicillin twice daily for five days.

Hypothesis

The proportion who fails treatment will be 10 percent in the reference group and the alternative treatment groups. An alternative therapy will be considered non-inferior to the standard therapy if the failure rate in the alternative therapy exceeds the failure rate in the injectable therapy by less than 5 absolute percentage points.

Secondary Objectives:

* To identify baseline clinical predictors of treatment failure in severe infections in young infants.
* To determine the proportion of relapse (young infants who were considered cured by day 7 but developed any of the signs of suspected severe infection by day 14).

DETAILED DESCRIPTION:
Although many developing countries have witnessed declines in both post-neonatal and 1-4 year-old child deaths, neonatal death rates have remained relatively constant, with an estimated 4 million annual neonatal deaths globally (Lawn et al, 2005). Almost all of the neonatal deaths (99%) occur in developing countries (Bryce et al., 2005; Ahmad et al., 2007). In many of these settings, the rate of home delivery is high and the attendance at birth by skilled personnel is low, leading to many babies being born in unhygienic conditions (Bhutta et al., 2005). Birth in these settings is accompanied by a high rate of infections in both mothers and newborns. It has been estimated that about 1 out of 5 neonates develop life threatening infections (Stoll, 1997). Several preventative interventions against neonatal infections including tetanus toxoid immunization to pregnant women, early and exclusive breastfeeding, and use of clean delivery kits have been identified and incorporated in many programs (Bhutta et al., 2005). Yet, neonatal infections remain the most important cause of neonatal deaths. Globally, an estimated one-third of the neonatal deaths are attributed to infections (Lawn 2005). In settings characterized by high neonatal mortality rates, the proportion of neonatal deaths due to infections has been estimated at approximately 50% (Bang 1999; Lawn 2005; Baqui 2006). These infectious deaths include sepsis, pneumonia, tetanus, meningitis and diarrhea. A further 27% of the neonatal deaths are related to premature birth and infections are the direct cause in many of these premature neonates. Therefore, strategies for timely identification and management of infections in young infants (0-59 days) including neonates are urgently needed.

Current Treatment Options: Hospital care The WHO recommends that all cases of suspected severe infection in young infants (0-59 days old) are treated in hospitals with a 7-10 day course of injectable antibiotics - penicillin (or ampicillin) and gentamicin. However, in many developing countries, this care is often not available or accessible, or not acceptable to families. Furthermore, in low-resource settings, reliance on a strategy of hospitalization of young infants with suspected severe infections has a number of inherent disadvantages. First, in many settings, a vast majority of young infants who are referred may not be able to get to the hospital (Peterson et al., 2004) and may not receive the treatment, increasing their risk of dying. Second, routine hospitalization and the use of injectable antibiotics, either intravenously or intramuscularly substantially increases the cost of health care (Al-Eidan et al., 1999) and often hospital beds are not available to admit all young infants with suspected serious infections. Third, hospitalization increases the risk of exposure to multi-drug resistant nosocomial pathogens that are increasingly difficult to treat (Jarvis WR, 2004; Pong et al., 2004).

Evidence of alternative approaches:

Strategies for community-based management of infections in young infants have been developed and evaluated in several research settings (Bang et al., 1999; Baqui et al., 2007; Kanal et al., 2007). Our group, known as Projahnmo, has recently completed a trial of a package of maternal and neonatal interventions in Sylhet district, Bangladesh, and demonstrated significant reduction of neonatal mortality (Baqui et al., 2008b). In one of the intervention arms, we trained village-based community health workers to assess newborns and manage newborns with severe infections using an algorithm similar to the one used in Integrated Management of Childhood and Neonatal Illness (IMNCI). Management included referral of neonates with signs of severe infection to a qualified provider and home treatment in referral failure cases. If referral failed but parents consented to home treatment, CHWs treated neonates with severe infections using injectable procaine penicillin and gentamicin. For severe infections, the rate of referral compliance was only 34%, and home treatment acceptance was 43%. The case fatality rate was 4.4% for those treated by CHWs, 14.2% for those treated by qualified medical providers, and 28.5% for those who either received no treatment or who were treated by untrained providers. After controlling for differences in background characteristics and illness signs among treatment groups, newborns treated by CHWs had a hazard ratio of 0.22 (95% confidence interval 0.07-0.71) for death during neonatal period and those treated by qualified providers had a hazards ratio of 0.60 (95% confidence interval of 0.37-0.99), compared to newborns who received no treatment or were treated by untrained providers (Baqui et al., 2007; Baqui et al., 2008a). These data suggest that treatment of neonates by CHWs was generally acceptable to the community. Home treatment of suspected sepsis in neonates by CHWs is effective in low-resource settings.

There are, however, major challenges associated with current community-based strategies for injectable therapy. First, it is difficult to ensure availability of trained health workers who are able to safely and optimally administer injectable antibiotics daily for 7 to 10 days, and to ensure supplies and quality assurance. Second, a 7 to 10-day regimen of parenteral antibiotic therapy presents specific challenges to community acceptance and compliance. Third, unsupervised use of injection at the community level may be unsafe and can increase the risk of transmission of HIV, hepatitis and other viral diseases through the use of contaminated needles (Simonsen et al., 1999). Therefore, it is important to reduce the number of injections to be used in the community. Furthermore, the rationale for 7-10 days of parenteral antibiotic therapy is not fully established. Injectable therapy is chosen because of the perception that it is the most efficacious regimen in the treatment of severe disease. For some neonatal infections, however, alternative regimes such as a combination of parenteral and oral therapy or switching to an oral antibiotic after initial treatment for 2-3 days with injectable antibiotics may be equally effective.

To overcome the disadvantages of hospitalization and challenges of community-based injectable therapy, recent research has looked at the potential use of oral treatment for severe pneumonia in older infants. Hazir et al (2008) recently reported the results from an open-label equivalency trial conducted at seven study sites in Pakistan. 2,037 children aged 3-59 months with severe pneumonia were randomly allocated to either initial hospitalization and parenteral ampicillin (100 mg/kg per day in four doses) for 48 h, followed by 3 days of oral amoxicillin (80-90 mg/kg per day in two doses; n=1012) or to home-based treatment for 5 days with oral amoxicillin (80-90 mg/kg per day in two doses; n=1025). Follow-up assessments were done at days 1, 3, 6, and 14 after enrolment. There was no difference in treatment failure rates (clinical deterioration) by day 7 between the hospitalized (8.6%) and the ambulatory group (7.5%; risk difference 1•1%; 95% CI -1•3 to 3•5). This result suggests empowering first-level health workers to manage severely ill children when referral is difficult. High failure rates were associated with young age, very fast breathing, and low weight for age. These findings suggest that it may not be safe to treat young infants with suspected severe infection with oral antibiotic alone.

Global research priority: Simplified antibiotic regimen for infections in young infants

In the fall of 2007, Saving Newborn Lives (SNL) of Save the Children-US, USAID and WHO convened a global consultation to review the new study findings on infection management in young infants in community-based settings and to guide future research priorities. Based on the existing research findings at that time, the consultation participants concluded that there was still insufficient evidence to make policy recommendations for global programs. The consultation charged future research to test optimal combination of oral and intramuscular (IM) antibiotic regimens that would be feasible to implement in first-level facilities and community and will be acceptable to families for settings characterized by weak health systems. We designed this study with these recommendations in mind.

ELIGIBILITY:
Inclusion Criteria:

* Infants 0-59 days old who are residents of catchment population of the study hospitals
* One or more of the following five signs: severe chest in-drawing, axillary temperature >37.80C or <35.50 C, lethargic or less than normal movement, and history of feeding problems (confirmed by poor suck on feeding assessment)
* Family refuses recommended hospitalization or hospitalization otherwise not feasible
* Informed consent by a legal guardian.

Exclusion Criteria:

* Very severe infection/disease characterized by presence of any of the following signs (unconscious, convulsions, unable to feed, apnea, unable to cry, cyanosis, bulging fontanel, major congenital malformations, major bleeding, surgical conditions needing hospital referral, persistent vomiting defined as vomiting following three attempts to feed the baby within ½ hour, and/or physician's suspicion of meningitis)
* Very low birth weight: weight <1500
* Hospitalization for illness in the last two weeks
* Hospital born infants
* Previous inclusion in the study

Max Age: 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2490 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Treatment failure | Seven days

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah H Baqui, MBBSMPHDrPH, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (3):
- Bangladesh (3):
  - Dhaka Shishu Hospital/CHRF, Dhaka, Dhaka Division
  - Chittagong Ma O Shishu Hospital, Chittagong
  - Shishu Shastya Foundation, Dhaka

REFERENCES:
- [Derived] Longombe AL, Ayede AI, Marete I, Mir F, Ejembi CL, Shahidullah M, Adejuyigbe EA, Wammanda RD, Tshefu A, Esamai F, Zaidi AK, Baqui AH, Cousens S. Oral amoxicillin plus gentamicin regimens may be superior to the procaine-penicillin plus gentamicin regimens for treatment of young infants with possible serious bacterial infection when referral is not feasible: Pooled analysis from three trials in Africa and Asia. J Glob Health. 2022 Nov 21;12:04084. doi: 10.7189/jogh.12.04084. PMID 36403158
- [Derived] Baqui AH, Saha SK, Ahmed AS, Shahidullah M, Quasem I, Roth DE, Samsuzzaman AK, Ahmed W, Tabib SM, Mitra DK, Begum N, Islam M, Mahmud A, Rahman MH, Moin MI, Mullany LC, Cousens S, El Arifeen S, Wall S, Brandes N, Santosham M, Black RE; Projahnmo Study Group in Bangladesh. Safety and efficacy of alternative antibiotic regimens compared with 7 day injectable procaine benzylpenicillin and gentamicin for outpatient treatment of neonates and young infants with clinical signs of severe infection when referral is not possible: a randomised, open-label, equivalence trial. Lancet Glob Health. 2015 May;3(5):e279-87. doi: 10.1016/S2214-109X(14)70347-X. Epub 2015 Apr 1. PMID 25841891
- [Derived] Baqui AH, Saha SK, Ahmed AS, Shahidullah M, Quasem I, Roth DE, Williams EK, Mitra D, Shamsuzzaman AK, Ahmed W, Mullany LC, Cousens S, Wall S, Brandes N, Black RE. Safety and efficacy of simplified antibiotic regimens for outpatient treatment of serious infection in neonates and young infants 0-59 days of age in Bangladesh: design of a randomized controlled trial. Pediatr Infect Dis J. 2013 Sep;32 Suppl 1(Suppl 1 Innovative Treatment Regimens for Severe Infections in Young Infants):S12-8. doi: 10.1097/INF.0b013e31829ff790. PMID 23945570